CLINICAL TRIAL: NCT04218409
Title: Opioid-Sparing and Pain-Reducing Properties of Syntocinon: A Dose-Effect Determination
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201902618-N; OCR30384 (Other: UF OnCore); 1K01DA052673-01A1 (NIH)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Oxycodone; Tablets

STUDY DESIGN:
Intervention Model Description: This is a within-participant study so that each participant receives all conditions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- oxycodone (5mg) + intranasal oxytocin (48 IU) (Active Comparator): Combined effects of oxycodone and oxytocin
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Oxytocin nasal spray
- Oral oxycodone (5mg) + intranasal placebo (Active Comparator): Separate effects of oxycodone. As is standard methodology in abuse liability and pain assessments a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Other: Placebo oxytocin
- oxytocin+placebo (Active Comparator): Separate effects of oxytocin. As is standard methodology in abuse liability and pain assessments a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo Oxycodone
- placebo+placebo (Sham Comparator): Serves as the control
  Interventions: Other: Placebo Oxycodone; Other: Placebo oxytocin
- Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU) (Active Comparator): Combined effects of oxycodone and oxytocin
  Interventions: Drug: Oxytocin nasal spray; Drug: OxyCODONE 2.5 mg Oral Tablet
- Oral oxycodone (2.5mg) + intranasal placebo (Active Comparator): Separate effects of oxycodone. As is standard methodology in abuse liability and pain assessments a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo
  Interventions: Other: Placebo oxytocin; Drug: OxyCODONE 2.5 mg Oral Tablet

INTERVENTIONS:
Drug: OxyCODONE 5 mg Oral Tablet — Oral oxycodone 5 mg orally
  Arms: Oral oxycodone (5mg) + intranasal placebo; oxycodone (5mg) + intranasal oxytocin (48 IU)
Drug: Oxytocin nasal spray — Intranasal oxytocin administration (48 IU)
  Arms: Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU); oxycodone (5mg) + intranasal oxytocin (48 IU); oxytocin+placebo
Other: Placebo Oxycodone — Oxycodone 0 mg orally
  Arms: oxytocin+placebo; placebo+placebo
Other: Placebo oxytocin — Intranasal placebo administration
  Arms: Oral oxycodone (2.5mg) + intranasal placebo; Oral oxycodone (5mg) + intranasal placebo; placebo+placebo
Drug: OxyCODONE 2.5 mg Oral Tablet — Oral oxycodone 2.5 mg orally
  Arms: Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU); Oral oxycodone (2.5mg) + intranasal placebo

SUMMARY:
Some research suggests that administration of oxytocin with oxycodone may reduce its abuse liability and improve its ability to reduce pain. In a 6-session laboratory study, the investigators will be evaluating the effects of oxycodone and oxytocin (combined and separately, across sessions) on experimentally-induced pain, subjective effects, decision-making, and activation of different neural substrates.

DETAILED DESCRIPTION:
The overall project goals are to determine oxytocin effects on oxycodone's subject-rated abuse liability, experimental pain, and to describe the neurobehavioral mechanisms underlying interindividual differences in these effects. Generally healthy individuals (determined via medical history review and a screening session) will, after informed consent, self-administer intranasal oxytocin (or placebo, containing the same ingredients but no oxytocin) shortly after oral oxycodone or placebo in a non-residential, double-blind, randomized, placebo-controlled, within-subjects laboratory study. Prescreening will assure MRI eligibility and drug application safety and, using a validated, comprehensive pain history interview, determine previous or existing chronic pain conditions, including current pain medication use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals fluent in English will participate.
* Must report recreational use of opioids.
* Be within 20% of their ideal body weight.
* Are not currently experiencing chronic pain (pain on most days during the past 3 months)
* Have a systolic blood pressure of <=140 and diastolic blood pressure of <= 90, and a heart rate <= 90 beats per minute.
* Participants must also have a normal electrocardiogram (EKG) reading and bloodwork indicating no major health contraindications.

Exclusion criteria:

* Significant current physical disease or major psychiatric disorder.
* No self-reported current interest in drug abuse treatment.
* Women who are pregnant or nursing.
* Any comorbid illicit substance use disorders or current clinically significant withdrawal for any abused drug excluding nicotine and caffeine.
* Any conditions that preclude safety in the MRI scanner, such as: implanted electrical devices (e.g., cardiac pacemaker, neurostimulator); implanted metallic clips or pins (e.g., aneurysm clip); a history of working with metal (unless able to demonstrate participant is MRI safe), and claustrophobia.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Subject-rated abuse liability | up to 6 weeks.
  Using a Visual Analog Scale with scoring as 0=not at all, 20=possibly mild, 40=definitely mild, 60=moderately, 80=strongly, and 100=extremely, or any number in between. Testing occurs only in the context of 4 sessions due to a minimum of a one week washout period in between each session.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Berry, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No